CLINICAL TRIAL: NCT05072028
Title: A Clinical Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]DBPR108 in Chinese Healthy Adult Male Subjects- Mass Balance and Biotransformation Study of [14C]DBPR108 in Human
Brief Title: Mass Balance and Biotransformation Study of [14C]DBPR108 in Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA1118-CSP-011
Record Dates: First submitted 2021-09-29; First posted 2021-10-08 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-09

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]DBPR108 (Experimental): Subjects will receive a single oral 100 mg (radioactivity of 150 µCi) dose of [14C]DBPR108 on Day 1.
  Interventions: Drug: [14C]DBPR108

INTERVENTIONS:
Drug: [14C]DBPR108 — [14C]DBPR108, single dose of 100 mg (radioactivity of 150 µCi), oral

SUMMARY:
This is a single-center, open-label phase I clinical study to evaluate the mass balance and biotransformation pathways of [14C]DBPR108 in Chinese healthy adult male subjects, to reveal the overall pharmacokinetic characteristics of DBPR108 in human body, and to provide a reference for the rational administration.

DETAILED DESCRIPTION:
This study will evaluate the mass balance and pharmacokinetics of DBPR108 in approximately 6 healthy male subjects receiving a single oral 100 mg dose of DBPR108 containing approximately 150 µCi of [14C]- DBPR108. This study consists of a screening period (Day -7 to Day -2), a baseline period (Day -1), a treatment period, and a follow-up visit period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults;
2. 18 to 45 years (inclusive);
3. Subjects weight ≥50.0 kg and body mass index (BMI) between18-26 kg/m^2 (inclusive) (BMI= weight (kg)/height^2 (m^2);
4. Medical history, vital signs examination, physical examination, laboratory tests (blood routine, blood biochemistry, urine routine, thyroid function) and other test results of subjects judged to be normal or abnormal without clinical significance;
5. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions.

Exclusion Criteria:

1. Clinically significant abnormal results for physical examination, vital signs, routine laboratory tests (blood routine, blood biochemistry, coagulation routine, urine routine, stool routine + occult blood, thyroid function, glycated hemoglobin), 12-lead electrocardiogram (ECG), chest CT scan, and abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, and kidney);
2. Any positive test result of hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
3. Subjects with a history of severe hypoglycemia, such as drowsiness, disturbance of consciousness, or even coma due to hypoglycemia;
4. History of acute and chronic pancreatitis, or a history of cholecystitis, gallstones, and pancreatic injury and other high-risk factors that may cause pancreatitis;
5. Subjects are hard to swallow, or have diseases affecting drug absorption, distribution, metabolism, excretion;
6. History of gastrointestinal ulcer or bleeding;
7. History of any clinically significant diseases, such as circulatory, endocrine, neurological, gastrointestinal, urinary, hematological, immunological, psychiatric and metabolic diseases;
8. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsade de pointes ventricular tachycardia, ventricular tachycardia, prolonged QT syndrome, or symptoms of prolonged QT syndrome and family history;
9. Have a major surgery or incomplete incision healing within 6 months prior to screening. Major surgery includes, but is not limited to, any surgery involving a significant risk of bleeding, prolonged general anesthesia, or open biopsy or obvious traumatic injury;
10. History of needle sickness or blood sickness, difficulty in blood collection or intolerance to venipuncture blood collection;
11. Have hemorrhoids or perianal disease with regular/ongoing bleeding stools;
12. Have habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease;
13. Have a history of allergic conditions, or have a history of allergy to any of DBPR108 or other similarly structured drugs. Those who cannot follow a uniform diet.
14. Subjects are lactose intolerant or have rare genetic galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption;
15. Use of any metabolizing enzyme inducers or inhibitors within 30 days prior to screening;
16. Use of any prescription drug, over-the-counter drug, proprietary Chinese medicine, herbal medicine, vitamins and supplements within 2 weeks prior to screening;
17. Have been vaccinated within 4 weeks prior to screening or who have a scheduled vaccinated plan during the study period;
18. Participation in another clinical trial within 3 months before screening (whichever is administrated);
19. Average weekly intake of alcohol is more than 14 units alcohol (1 units ≈ 360 mL beer, or 45 mL spirits with 40% content, or 150 mL wine) within the 6 months prior to screening, or a positive ethanol breath test at screening;
20. Smoking more than 5 cigarettes per day within 3 months prior to screening, or who cannot stop using any tobacco products during the study period;
21. History of drug abuse, or positive urine drug screen at screening;
22. Subjects who have a habitual consumption of grapefruit juice or excessive amounts of tea, coffee and/or caffeinated beverages (such as coffee, tea, cola, chocolate, energy drinks), and unable to quit during the study period;
23. Workers engaged in long-term exposure to radioactive conditions, or have had significant radiation exposure (≥2 chest/abdominal CT scans, or ≥3 other types of X-rays) or participated in the radiopharmaceuticals labeling test within 1 year prior to the study;
24. Subjects who have fertility or sperm donation plans, or do not agree to use strict contraceptive methods during the study period and within 1 year after the completion of the study;
25. Blood donation (or blood loss) ≥400 mL within 3 months, or receiving whole blood transfusions or erythrocyte suspension transfusions within 1 month prior to the screening;
26. Not suitable for this study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in urine and feces | From time zero up to 240 hours post-dose following oral administration of [14] DBPR108
Peak plasma concentration (Cmax) | From time zero up to 96 hours post-dose following oral administration of [14] DBPR108
Area under the plasma concentration versus time curve from time zero to the last measurable concentration (AUClast) | From time zero up to 96 hours post-dose following oral administration of [14] DBPR108
Area under the plasma concentration versus time curve from time zero to infinity (AUCinf) | From time zero up to 96 hours post-dose following oral administration of [14] DBPR108
Time to achieve maximum plasma concentration (Tmax) | From time zero up to 96 hours post-dose following oral administration of [14] DBPR108

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed by CTCAE v5.0 | From time zero up to 240 hours post-dose following oral administration of [14] DBPR108

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, China